CLINICAL TRIAL: NCT02705690
Title: Benchmarking the iOS Balance Application Against the Berg Balance Test
Acronym: BBAaBBT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Stannah Stairlifts (Industry)
Collaborators: University College, London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Stannah_Balance_01
Record Dates: First submitted 2016-03-07; First posted 2016-03-10 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Arthroplasty, Replacement, Hip; Arthroplasty, Replacement, Knee; Ankle Injuries; Knee Injuries; Accidental Falls; Spinal Injuries
MeSH Terms: conditions — Ankle Injuries; Knee Injuries; Spinal Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: iOS Balance Application — We have designed an iOS application and a belt. The application uses accelerometer data to calculate postural sway. Steps:
  The phone is kept stable against the lower back of the participant using the belt.
  The iOS application gives instructions to user to adopt the correct stance (eg: Standing Unsupported, legs side by side) Once the stance is adopted, the application turns on the accelerometer in the phone to sample acceleration along x (media lateral) and z (anterior posterior) axis.
  These displacements from the mean are used to calculate the Root Mean Square of a person which acts a proxy score for Postural Sway. (Postural sway is defined as the phenomenon of constant displacement and correction of the position of the center of gravity within the base of support)

SUMMARY:
This study aims to benchmark the performance of an iOS application against the Berg Balance Scale (BBS), which is the most commonly used assessment tool by clinicians for measuring balance across the continuum from acute care to community-based care. An iPhone will be tied around the waist of the participant and concurrent measurements will be taken for five of the fourteen stances which comprise the BBS.

DETAILED DESCRIPTION:
'Project Balance' aims to make balance an actionable component of an individuals health, allowing a long term intervention via a monitoring and training of balance health much before a fall happens. Towards this end, we have designed an iOS application and a belt. The phone is kept stable against the lower back of the participant using the belt. The application turns on the accelerometer in the phone to sample acceleration along x (media lateral) and z (anterior posterior) axis. These displacements from the mean are used to calculate the Root Mean Square of a person which acts a proxy score for Postural Sway. (Postural sway is defined as the phenomenon of constant displacement and correction of the position of the center of gravity within the base of support)

Studies in the past have compared the use of accelerometers to the use of the clinical measured of Timed Up (TUG) test and Berg Balance Scale (BBS) in the assessment of postural stability and indicated that there is a high correlation between BBS, TUG and Accelerometry. Accelerometry has also found to be able to distinguish between sway responses to differing balancing conditions and between fallers and non-fallers.

We aim to conduct a benchmarking study for our iOS application against the BBS.

ELIGIBILITY:
Inclusion Criteria:

Between the ages of 18 - 69 Selected to undergo a Berg Balance Sale Impairments including : Ankle injures, Knee Replacements, Hip Replacements, Knee injuries, ligament tears etc.

Exclusion Criteria:

Subjects will be excluded from participation if they have peripheral neuropathy (clinically diagnosed or if they had symptoms of numbness/tingling in the lower extremities); pain of any level presenting simultaneously in both lower extremities; or unilateral lower extremity pain >3 on the 11 point visual analog (box) scale. Pregnant women will be excluded.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-06 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Spearman's Rank Coefficient to compare the Root Mean Square from iOS application to the Berg Balance Scale Score | Baseline

SECONDARY OUTCOMES:
Symmetry Ratio (Root Mean Square Left Leg vs Root Mean Square Right Leg) AP/ML Ratio (Ratio of the Anterior Posterior movement vs the media lateral movement) | Baseline
  The iOS application can compare the Root Mean Square(RMS) from the left leg to the right leg to produce a symmetry ratio for the physiotherapist, this provides a more granular view of the participants balance health. Similarly, the application can calculate the ratio of Anterior Posterior movement to the Media Lateral movement.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Prince Charles Hospital, Gurnos Rd, Merthyr Tydfil
  - Prince Charles Hospital, Cardiff